CLINICAL TRIAL: NCT05019365
Title: Investigating the Long-term Cardiac Sequelae of Trastuzumab Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other); Tenovus Scotland (Other)
Responsible Party: Principal Investigator, Kenneth Mangion, Principal Investigator, University of Glasgow
Other Study IDs: GN19ON381
Record Dates: First submitted 2020-11-24; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer; Cardiotoxicity
Keywords: Cardiotoxicity; HER2-positive Breast Cancer; Cardiac MRI
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with previous HER2 breast cancer
- Healthy Volunteers

SUMMARY:
The introduction of trastuzumab for the treatment of patients with human epidermal growth factor receptor 2 (HER2) positive breast cancer has had a major impact upon cancer outcomes. However, cardiac toxicity remains a substantial concern. Conventionally, this toxicity has been considered as a transient and reversible phenomenon occurring in the immediate peri-treatment period in around 20% of patients. Current guidelines recommend monitoring heart function during treatment and at completion. Recent registry data suggest that trastuzumab-related cardiotoxicity may also manifest in the longer-term. The nature and longer-term prevalence of left ventricular dysfunction with HER2 positive breast cancer treated with trastuzumab is unclear. The aim of this project is to define the prevalence of left ventricular dysfunction late after completion of trastuzumab therapy.

DETAILED DESCRIPTION:
In 2014, there were 45,535 cases of breast cancer diagnosed in England and Wales(1). Predicted 10-year survival in 2015, from data by the National Statistics office was estimated at 81%(2). Breast cancer is the most common malignancy in Scotland and the second most common cause of death(3). Around 1 in 4 of these cancers overexpress human epidermal growth factor receptor 2 (HER2). For these patients, trastuzumab is a recommended and highly effective component of a chemotherapy regime that usually includes an anthracycline(4).

Up to a quarter of patients treated with trastuzumab will develop cardiac dysfunction(5-7), conventionally defined as an asymptomatic >10% fall in left ventricular ejection fraction (LVEF) to an absolute LVEF <50%, or symptomatic heart failure(8). The risk is greater in patients who have received prior anthracyclines(9). Trastuzumab-related cardiotoxicity has, typically been considered to be a reversible phenomenon which recovers with interruption or cessation of treatment(10-14). The long-term benefit of cardioprotective treatment with angiotensin converting enzyme inhibitors or beta blockers when cardiotoxicity is detected is unclear(8) and these agents are often either not continued or not be prescribed at all.

The incidence of cardiac dysfunction or heart failure in the longer-term is not well-defined (12,14-20) . Clinical trials, which have excluded patients with baseline cardiovascular comorbidity, report no excess of cardiovascular events after the first two years(21-23) but observational studies report a much higher incidence of up to 23.8%(9,24). A landmark analysis of patients with a history of breast cancer (median follow-up 9 years) reported that patients treated with anthracycline chemotherapy and trastuzumab were three-fold more likely to develop heart failure than those treated with anthracycline alone. Importantly, these data were derived from a population censored at one year and reflect 'late' manifestations of cardiotoxicity rather than ongoing symptoms from an early diagnosis(25). This important study reported the incidence of symptomatic heart failure and not LV dysfunction which would be expected to be substantially more prevalent(26). Furthermore, the long-term implications of an apparently transient drop in LVEF during treatment are unclear.

Cardiovascular magnetic resonance (CMR) is the gold standard for the assessment of LV function(27). Previous work has demonstrated that CMR may be better able to identify small changes in LVEF related to chemotherapeutic agents(18,28,29). CMR has superior accuracy and precision when compared with echocardiography and allows myocardial tissue characterisation(30,31). My proposed CMR protocol will generate important insights into the long-term cardiac effects of trastuzumab and further novelty will be provided by the incorporation of tissue mapping methods(32) and LV strain assessment(33,34). Via collaboration with mathematicians I will also derive computational models.

ELIGIBILITY:
Inclusion Criteria:

* patients with HER2 positive breast cancer who received anthracycline-containing chemotherapy followed by trastuzumab at least 5 years prior to enrolment;
* age >18 years.

Exclusion Criteria:

* standard contraindication to CMR (ex: pacemaker, metallic implant);
* pregnancy;
* eGFR <30 ml/min/1.73 m2) past medical history of heart failure or left ventricular systolic dysfunction.

Healthy Volunteers:

Twenty age and sex matched healthy volunteers will undergo a similar CMR protocol.

Inclusion Criteria:

* least 18 years (they will be matched to the study participants)
* no prior medical history (including cardiovascular health problems, medication or systemic illness)

Exclusion Criteria:

* standard contraindication to CMR;
* suspected pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were treated with anthracycline and adjuvant trastuzumab chemotherapy at least 5 years previously.
  Age matched healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-05-25 (Estimated); Study Completion 2022-11-25 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Systolic Dysfunction | Through study completion, on average <2years.
  To define the prevalence of left ventricular dysfunction in patients who received trastuzumab chemotherapy at least 5 years previously
Reduced Global Longitudinal Strain (global and segmental) | Through study completion, on average <2years.
  GLS less than 2 standard deviations from normal reference range, using Displacement Encoding with Stimulated Echoes (DENSE) MRI.
Reduced Circumferential Strain (global and segmental) | Through study completion, on average <2years.
  GCS less than 2 standard deviations from normal reference range, using Displacement Encoding with Stimulated Echoes (DENSE) MRI.

OTHER OUTCOMES:
T1 relaxation times (global and segmental) | Through study completion, on average <2years.
  Left ventricular (LV) Parametric maps (T1, T2, Extracellular volume) will be assessed using a 16 segment model with bespoke MRI analysis software.
T2 decay time (global and segmental) | Through study completion, on average <2years.
  Left ventricular (LV) Parametric maps (T1, T2, Extracellular volume) will be assessed using a 16 segment model with bespoke MRI analysis software.
Extracellular volume fraction (ECV) (global and segmental) | Through study completion, on average <2years.
  Left ventricular (LV) Parametric maps (T1, T2, Extracellular volume) will be assessed using a 16 segment model with bespoke MRI analysis software.
Presence of scar by late gadolinium enhancement (LGE) | Through study completion, on average <2years.
  Late gadolinium enhancement will be assessed using a 16 segment model with bespoke MRI analysis software.
Aortic Stiffness | Through study completion, on average <2years.
  Aortic stiffness will be assessed using MRI sequences.
ECG abnormalities | Through study completion, on average <2years.
  Rhythm and heart rate will be recorded. Evidence of LVH, ST segment deviations and T wave flattening/inversion, and conduction abnormalities including QRS and QT interval will be recorded.
Computational Modelling | Through study completion, on average <2years.
  To identify novel biomarkers of heart pump function through the generation of computational models in patients who received trastuzumab and age matched healthy volunteers.

CONTACTS AND LOCATIONS:
Locations (1):
- Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will be on reasonable request to CI.